CLINICAL TRIAL: NCT04069325
Title: Efficacy and Safety of Simiaowan in Prevention of Acute Flares in Chronic Gout Patients Initiating Febuxostat Therapy：a Randomized Controlled Trial
Brief Title: Efficacy and Safety of Simiaowan in Prevention of Acute Flares in Chronic Gout Patients Initiating Febuxostat Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Affiliated Hospital of Nanjing University of Chinese Medicine (Other); The Second Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Principal Investigator, Quan Jiang, Director, Devision of Rheumatology, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: WD-18-F02
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Gout Flare
Keywords: gout; acute flares; prevention; febuxostat
MeSH Terms: conditions — Gout | interventions — simiaowan; Febuxostat

STUDY DESIGN:
Intervention Model Description: 72 subjects will be randomized to two parallel groups (36 subjects per group) to receive simiaowan 6g twice daily or placebo. All subjects will be given febuxostat 40mg once daily as background therapy. Placebo will be administered to individuals randomized to that treatment group in a form identical to the simiaowan. The first investigational medicinal product dose will be administered the day after the randomization.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- simiaowan 6g + febuxostat 40mg (Experimental)
  Interventions: Drug: simiaowan; Drug: febuxostat
- placebo 6g + febuxostat 40mg (Placebo Comparator)
  Interventions: Drug: placebo; Drug: febuxostat

INTERVENTIONS:
Drug: simiaowan — pills, 6g twice daily (BID), oral, 12 weeks
  Arms: simiaowan 6g + febuxostat 40mg
Drug: placebo — pills, 6g twice daily (BID), oral, 12 weeks
  Arms: placebo 6g + febuxostat 40mg
Drug: febuxostat — tablets, 40 mg once daily (QD), oral, 12 weeks

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of simiaowan in prevention of acute flares in chronic gout patients initiating febuxostat therapy.

DETAILED DESCRIPTION:
The study is a multicenter, randomized, double-blind, placebo-controlled, 12-week trial. To determine whether oral simiaowan at standard clinical doses (6g twice daily), compared to placebo, can reduce the incidence of acute gout flares and decrease the serum uric acid level.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 to 75 years (time of get informed consent)
* Meet the American College of Rheumatology/The European League Against Rheumatism criteria (2015) for the classification of acute arthritis of primary gout
* Pain Visual Analogue Scale Score (VAS) ≤ 3 at screening
* Serum uric acid ≥7 mg/dL (420μmol/L) at screening
* Self-reported history of at least 2 gout flares within 12 months prior to screening
* Normal electrocardiogram (ECG), or no clinical significant at screening
* Be capable of understanding and complying with protocol requirements

Exclusion Criteria:

* Occurrence of an acute gout flare ongoing at screening or within 2 weeks prior to screening
* Known or suspected of secondary hyperuricemia (e.g. due to renal disorder, hematological disorder, drugs, radiotherapy, chemotherapy or organ transplant)
* Use of colchicine, allopurinol, probenecid, benzbromarone, febuxostat or history of intra-articular steroid injection within 4 weeks prior to screening
* Use of glucocorticoids, nonsteroidal antiinflammatory drugs (NSAIDs), or cyclooxygenase-2 (COX-2) inhibitors within 1 week prior to screening
* History of stroke, transient ischemic attack (TIA), acute myocardial infarction (MI), heart failure (NYHA Class II-IV), coronary intervention procedure (including but not limited to angioplasty, stent placement, coronary revascularization) prior to screening
* History of gastrointestinal (GI) bleeding, peptic ulcer disease prior to screening
* History of malignancy and/or mental disorder prior to screening
* Active infection with hepatitis B, hepatitis C, or has aspartate transaminase (AST), alanine aminotransferase (ALT) or gamma-glutamyl transpeptidase (GGT) values ≥1.2 times the upper limit of normal (×ULN) during the screening period
* Presence of severe renal function impairment, or has serum creatinine (sCr) values ≥1.2 (×ULN) during the screening period
* History of allergy or intolerance to febuxostat, diclofenac sodium, simiaowan and/or the placebo
* History of aspirin-induced asthma, or any other form of allergy to aspirin and other NSAIDs
* Other (non-gout) chronic arthritis, acute inflammatory arthritis, autoimmune diseases with arthritis at screening
* Being treated with simiaowan at screening
* Being treated with azathioprine, mercaptopurine, theophylline, cytotoxic agents at screening
* Diagnosis of drug or alcohol dependence or abuse or any condition requiring chronic daily use of pain medication
* Pregnant or nursing, or planning to become pregnant or father a child within 3 months after receiving the last dose of study drug
* Subjects who participated in another clinical study or clinical trial within 3 months prior to screening
* Any other condition(s) that will compromise the safety of the patient, prevent compliance with the study protocol, or compromise the quality of the clinical study, as judged by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-07-28 (Estimated); Study Completion 2020-07-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects experiencing ≥ 1 gout flare within 12 weeks | Day 1 to Week 12
  Proportion of subjects in each group who experiencing at least 1 new gout flare during the 12 weeks study treatment period.

SECONDARY OUTCOMES:
The incidence of new gout flares within 12 weeks in the simiaowan group compared to the placebo group | Day 1 to Week 12
  For each new flare, subjects will be asked to record in their patient diary. The total incidence of new gout flares is reported during the 12-week study treatment period.
Proportion of subjects in each group achieving serum uric acid concentration≤ 7 mg/dL (420μmol/L) | Week4, Week 8 and Week 12
Proportion of subjects experiencing from ≥ 1 gout flare and ≥ 2 gout flares within 12 weeks | Day 1 to Week 12
Mean pain Visual Analogue Scale Score (VAS) associated with gout flares | Day 1 to Week 12
  Subjects who experience an acute gout flare within 12 weeks will be asked to score their pain intensity in the most affected joint on a 0-10 mm Visual Analogue Scale Score (VAS), ranging from no pain (0) to extremely pain (10).
Amount of rescue medication taken within 12 weeks | Day 1 to Week 12
  Subjects who have difficulty in tolerating the pain of an acute gout flare will be allowed to take rescue medication (diclofenac sodium, 25mg, three times daily).

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Quan, Doctor, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No